CLINICAL TRIAL: NCT05819606
Title: PERsonalized Positron Emission Radiomics With Prostate Cancer Specific Membrane Antigen Radioligands on Newly Diagnosed Prostate Cancer Patients.
Brief Title: Positron Emission Radiomics With PSMA Radioligands on Newly Diagnosed Prostate Cancer Patients
Acronym: PER2PSMA
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5641
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Immunohistochemistry (IHC) analysis — Setting of the percentage amount of PSMA expression on the primary tumor cell surface on post-surgical samples by the Immunohistochemistry method (IHC)

SUMMARY:
The primary aim of this large prospective study consists of exploring the correlation among Volumetric and Radiomic parameters extracted from staging PSMA PET/CT Imaging versus conventional baseline clinical biochemical data, conventional imaging and the aggressiveness of the tumor based on the post-surgical-Gleason Score (GS) in patients with intermediate/high risk prostate cancer (PCa).

Secondarily, Volumetric and Radiomic features extracted from the same PET images will be compared with the amount of the Circulating Tumor Cells (CTCs), with the expression of specific receptors on CTCs surface,

Possible mutations encoding androgen receptors (AR) on CTCs surface, and with PSMA density on primary tumor cells provided by the Immunohistochemistry method (IHC) applied on post-surgical histological samples.

According to PET images, Volumes of interest (VOI) encompassing the whole prostate with foci of PSMA uptake suspected for PCa will be drawn to extract semiquantitative and radiomic PET features.

The association between PSMA PET radiomics and CTCs molecular and genomic panel at staging could potentially lead to a more personalized and more effective therapeutic chances.

DETAILED DESCRIPTION:
The following clinical conventional parameters will be collected :

* age (years),
* results of DRE, digital rectal examination (positivie or negative)
* Prostate-Specific Antigen. PSA levels (ng/ml)
* conventional PET parameters and ,(tSUVmax, tSUVmean, tMTV, tTLA),
* first-order radiomic features (tSkewness, tKurtosis)
* results from mpMRI (PIRADS categories from 1 to 5 according to v2.1)
* biopsy-based Gleason Score, GS (referrred to WHO/ISUP score)
* the amount of circulating tumor cells by the bloodstream peripheral samples CTCs (cells number/ml of blood volume)
* the overexpression of specific receptors on the CTCs surface, such as the epidermal grow factor receptor (EGFR), PSMA receptor.
* percentage of expression of specific receptors and their potential mutations on CTCs surface, in terms of percentage of expression of PSMA and GRPR based on histological post-surgical specimen on tumor cell surface.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign informed consent
* Biopsy-confirmed intermediate/high risk prostate cancer
* Good compliance to undergo mpMRI scan and PET/CT scan
* Eligible for radical prostatectomy

Exclusion Criteria:

* Contraindication to mpMRI (such. Metal implants and/or pacemaker)
* Poor compliance to undergo PET/CT (i.e.claustrophobia)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed biopsy confirmed intermediate/high risk PCa will be consecutively enrolled.
  All patients will undergo a multiparametric MRI (mpMRI) examination at Radiology Department and a PET/CT with PSMA radioligands for staging in the PET/CT Center, both in the Fondazione Policlinico Universitario A. Gemelli IRCCS (Rome, Italy). After PET scan all patients will be eligible for radical prostatectomy.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of aggressiveness of prostate cancer. | 9 months
  Prostate cancer evaluation of aggressivness via semiquantitative and volumetric PSAM PET features

SECONDARY OUTCOMES:
Radiogenomic panel of prostate cancer. | 9 months
  CTCs correlation with Prostate cancer aggressivness expressed by Gleason Score

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Annunziata, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- GSTeP FPG Policlinico Gemelli IRCCS, Roma, Italy